CLINICAL TRIAL: NCT01311401
Title: Predictors of Future Type 2 Diabetes Mellitus in Circassians Minority in Israel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Collaborators: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Osamah Hussein, Dr. Osamah Hussein, Ziv Hospital
Other Study IDs: 0067-08
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus Type II
Keywords: 2 diabetes mellitus,Circassians, High fasting glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rehania village (Kfar Rehania): Circassian community
  Interventions: Other: NONE intervention
- Kama village (Kfar Kama ): Circassian community
  Interventions: Other: NONE intervention

INTERVENTIONS:
Other: NONE intervention — NONE intervention

SUMMARY:
The aim

The aim of the present study is:

1. The metabolic risk factors that can predict diabetes after 10 years in a Circassians population-based sample of people who were aged 35 years or older and living in Israel.
2. To define the incidence of type 2 diabetes mellitus in Circassians minority in Israel.

The hypothesis of the study:

High fasting glucose has the most powerful predictive value for type 2 diabetes mellitus in the future.

The claimed importance of the study:

Finding a powerful risk factor for future diabetes mellitus can contribute to intensifying the preventive measures in a small part of the population, by that to reduce the incidence of new diabetes without increasing the health cost.

DETAILED DESCRIPTION:
Research design and methods The present study is a 10 year, nested prospective cohort, population-based survey of the metabolic syndrome risk factors including type 2 diabetes mellitus. The original cross-sectional survey was conducted in two small Circassian villages in north Israel with 4000 inhabitants. The baseline evaluation was performed between 1996 and - 1997. Among the 739 randomly selected men (n=289) and women (n=450 of the 4000 individuals who were aged 35 years or older. Mean age of men was 53.2±11.8 years and of women was 52± years. Mean BMI for men and women was 27.5± and 29.4± Kg/m2, respectively. Plasma glucose level for men and women was mg/dL(22).

The investigators will recruit the same cohort in the proposed study and individuals who were free of diabetes at base line will be included. The number of deceased changed their residence and those who will decline to participate in the follow-up study will be reported.

The protocol was approved by the Ethics Committee of the Ziv hospital and all participants will give an informed consent.

Clinical data. Body mass index (BMI), fasting blood glucose, blood total cholesterol, triglycerides, low density cholesterol (LDL), high density cholesterol (HDL) and blood pressure measurements were done 10 years ago. In the present study, after 8 hours of caloric fast, blood glucose levels will be tested and patients will be asked about known recent diabetes mellitus in the last 10 years or treatment by dietary, hypoglycemic drugs or insulin.

Laboratory data. In the morning, after an overnight caloric fast, venous blood will be sampled for the measurement of plasma concentrations of glucose. The blood levels of glucose will be done by Olympus 640 at ZIV hospital. Diagnosis of diabetes. At baseline and at the 10-year follow-up, the presence of diabetes will be established according to World Health Organization (WHO) criteria (84), i.e., when fasting glucose will be ≥126 mg/dl or when the participants will have a clinical diagnosis of the disease and treatment was ongoing (diet, drugs).

The presence of the disease will be confirmed by reviewing the medical records of their general practitioners. No case of diabetes will be accepted without a validated confirmation.

ELIGIBILITY:
Inclusion Criteria:

Previous participation in similar study which was occured 10 years ago

Exclusion Criteria:

none

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Circassians in Israel
Sampling Method: Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2009-10; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
New incidences of Type II Diabetes Mellitus in Circassians minority in Israel | 14 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel